CLINICAL TRIAL: NCT02978677
Title: Proton Dose Escalation for Patients With Atypical or Anaplastic Meningiomas
Acronym: PANAMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Cancer Research Center (Other); Radiation Oncology Working Group of the German Cancer Society (Other)
Responsible Party: Principal Investigator, Mechthild Krause, Principal Investigator, Technische Universität Dresden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STR-PANAMA-2015
Record Dates: First submitted 2016-10-19; First posted 2016-12-01 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Meningioma
Keywords: brain tumors; proton radiotherapy; photon radiotherapy
MeSH Terms: conditions — Meningioma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grade II tumors (macroscopic) (Experimental): Radiotherapy 68 Gy(RBE)
  Interventions: Radiation: Radiotherapy 68 Gy(RBE)
- Grade III tumors (macroscopic) (Experimental): Radiotherapy 72 Gy(RBE)
  Interventions: Radiation: Radiotherapy 72 Gy(RBE)
- Grade II/III tumors (completely resected) (Active Comparator): Radiotherapy 60 Gy(RBE)
  Interventions: Radiation: Radiotherapy 60 Gy(RBE)

INTERVENTIONS:
Radiation: Radiotherapy 68 Gy(RBE) — Radiotherapy 2.0 to 50 Gy(RBE) photon or proton and boost 2 to 18 Gy(RBE) proton
  Arms: Grade II tumors (macroscopic)
Radiation: Radiotherapy 72 Gy(RBE) — Radiotherapy 2.0 to 50 Gy(RBE) photon or proton and boost 2 to 18 Gy(RBE) proton and boost 2 to 4 Gy(RBE) proton
  Arms: Grade III tumors (macroscopic)
Radiation: Radiotherapy 60 Gy(RBE) — Radiotherapy 2.0 to 50 Gy(RBE) photon or proton and boost 2 to 10 Gy(RBE) proton
  Arms: Grade II/III tumors (completely resected)

SUMMARY:
The trial evaluates the effect of a moderately increased radiation dose in patients with atypical (grade II) and anaplastic (grade III) meningioma after incomplete or no surgery. Endpoint is recurrence-free survival after 5 years.

DETAILED DESCRIPTION:
The trial intends to optimize treatment for grade II and grade III (atypical or anaplastic) meningioma. Standard treatment for atypical or anaplastic meningioma is surgery. For grade III (anaplastic) meningiomas, post-operative radiotherapy would be performed in all cases using standard fractionation schedules to a total dose of ~60 Gy. For grade II (atypical) meningiomas, although some small patient datasets support early onset of radiotherapy, the standard treatment is still to irradiate if tumours are recurrent or if resection was macroscopically incomplete. Total doses of 54 to ~60 Gy are applied using standard fractionation schedules.

A major problem of the treatment of atypical or anaplastic meningioma is that beyond surgery and radiotherapy, there are only experimental treatment options and the probability of local recurrences is 50-100% within the first 5 years for grade II and grade III meningioma.

The present trial has been developed to evaluate efficacy of a dose-intensified radiotherapy treatment schedule for incompletely or not resected meningioma to a total dose of 68 (grade II) or 72 Gy (grade III). To minimize normal tissue toxicity, the boost dose or the complete radiotherapy is applied using protons. The expectation is a higher recurrence-free survival compared to previous reports on outcome of standard dose (60 Gy) radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed atypical (WHO grade II) or anaplastic (WHO grade III) meningioma with the indication for radiotherapy
* MRI (within 24h post-operative, if not available than with a time interval of ~ 6 weeks) including contrast-enhanced T1 weighted 3D dataset and PET for evaluation of macroscopic tumour (residuum)
* Karnofsky Performance Score ≥ 60, ECOG ≤2
* For women with childbearing potential, (and men) adequate contraception.
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* refusal of the patients to take part in the study
* previous radiotherapy of the brain
* several manifestations of the meningioma in different regions of the brain or additional spinal manifestations
* distant metastases
* patients who are not suitable for radiotherapy
* known other malignant disease within 5 years before radiotherapy (except tumours that likely do not impact prognosis and likely not require treatment interfering with study therapy, e.g. in-situ carcinoma of the breast or cervix uteri)
* pregnant or lactating women
* patients with non-MRI compatible metal implants, pacemaker or non-MRI compatible external automatic defibrillators
* patients not able to understand character and individual consequences of the clinical trial
* claustrophobic patients
* current participation in another clinical intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 5 years after start of radiotherapy

SECONDARY OUTCOMES:
late toxicity | 5 years after start of radiotherapy
  CTC-AE 4.0
acute toxicity | 5 years after start of radiotherapy
  CTC-AE 4.0
overall survival | 5 years after start of radiotherapy
patterns of recurrence using MRI | 5 years after start of radiotherapy
quality of life by validated quality of life questionnaires | 5 years after start of radiotherapy
  EORTC-QLQ-C30, EORTC-QLQ-BN20

CONTACTS AND LOCATIONS:
Overall Officials: Mechthild Krause, Prof., Study Chair — Technische Universität Dresden, German Cancer Consortium, Helmholtz-Zentrum Dresden - Rossendorf

IPD SHARING:
Plan to Share IPD: No